CLINICAL TRIAL: NCT04318652
Title: The Role of Anterior Segment Optical Coherence Tomography in Management of Acquired Punctal Stenosis
Brief Title: OCT Guided Punctal Stenosis Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Mahmoud Awara, assistant professor of ophthalmology, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32399/09/18
Record Dates: First submitted 2020-03-15; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Epiphora Due to Insufficient Drainage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone eye drops (Other): Preservative free steroids methylprednisolone 5% eye drops (prepared by dilution of methyleprednisolone 500mg in 10 ml distilled water (Solu-Medrol, Pfizer company) was prepared and given for all enrolled cases by the following regimen 5 times/day for 5 days with gradual decrease every third day over the following 2 weeks
  Interventions: Drug: Methylprednisolone eyedrops
- distilled water eyedrops (Placebo Comparator): Distilled water eyedrops instilled 3 times per day for two weeks
  Interventions: Drug: Methylprednisolone eyedrops

INTERVENTIONS:
Drug: Methylprednisolone eyedrops — instillation of methylprednisolone eye drops

SUMMARY:
This is a clinical trial study that was conducted on patients with punctal stenosis.We studied the diameter of stenosed puncta before and after treatment with preserved free steroid eye drops using AS-OCT.

DETAILED DESCRIPTION:
The study was conducted on 40 eyes of 24 patients have acquired inflammatory punctal stenosis and 20 eyes of 10 patients of normal asymptomatic subjects as control group. We studied the external punctal diameter, visibility of the internal punctum and punctal depth before treatment using AS-OCT, and then patients were re-evaluated after one month of treatment with preservative free methylprednisolone 5% eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Patients have acquired inflammatory punctum stenosis complaining of epiphora of different etiologies.

Exclusion Criteria:

* Previous lacrimal surgery.
* Lid margin malposition such as ectropion, entropion or lid retraction.
* Medial lid masses obscuring punctum.
* History of ocular trauma involving lid margin or punctum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
punctal opening | one month
  evaluation of punctalopening by OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Awara, Tanta, Gharbeyia, Egypt